CLINICAL TRIAL: NCT06622915
Title: Cardiac Performance Evaluation in Children With Steroid Dependent vs Steroid Resistant Nephrotic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa yahia Mohamed, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: soh_med_24_07_03MS
Record Dates: First submitted 2024-08-28; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A, (Active Comparator): steroid dependent nephrotic syndrome
  Interventions: Device: Tissue Doppler imaging and Conventional Echocardiography
- Group B (Active Comparator): steroid resistant nephrotic syndrome
  Interventions: Device: Tissue Doppler imaging and Conventional Echocardiography

INTERVENTIONS:
Device: Tissue Doppler imaging and Conventional Echocardiography — non-invasive cardiac imaging technique which measures the velocity of the longitudinal motion of the mitral annulus, tricuspid annulus and the basal part of interventricular septum
  Other Names: Conventional Echocardiography

SUMMARY:
nephrotic syndrome (NS) is one of the most common pediatric kidney diseases There is an increased incidence of heart disease in patients with primary nephrotic syndrome (PNS) compared to the normal population Conventional Echocardiography is usually utilized to diagnose myocardial dysfunction. Tissue Doppler imaging is a non-invasive cardiac imaging technique which measures the velocity of the longitudinal motion of the mitral annulus, tricuspid annulus and the basal part of interventricular septum

ELIGIBILITY:
Inclusion Criteria:

* Children with primary nephrotic syndrome.

  * Age: 2 - 14 years.
  * Both males and females

Exclusion Criteria:

* Patients of primary cardiac diseases (e.g., congenital or rheumatic heart disease, cardio- myopathy).

Patients who refuse to give written informed consent to study

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
cardiac performance evaluation in children with steroid dependent vs steroid resistant nephrotic syndrome | 12 months
  compairing of myocardial performance index (MPI)(Tei index) in nephrotic dependant and resistant nephrotic syndrom by calculating ejection time (ET) of right and left ventricle and mitral closure time (MCT) using tissue doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banh THM, Hussain-Shamsy N, Patel V, Vasilevska-Ristovska J, Borges K, Sibbald C, Lipszyc D, Brooke J, Geary D, Langlois V, Reddon M, Pearl R, Levin L, Piekut M, Licht CPB, Radhakrishnan S, Aitken-Menezes K, Harvey E, Hebert D, Piscione TD, Parekh RS. Ethnic Differences in Incidence and Outcomes of Childhood Nephrotic Syndrome. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1760-1768. doi: 10.2215/CJN.00380116. Epub 2016 Jul 21. PMID 27445165
- [Background] Correia Pinto J, Henriques-Coelho T, Roncon-Albuquerque R Jr, Leite-Moreira AF. Differential right and left ventricular diastolic tolerance to acute afterload and NCX gene expression in Wistar rats. Physiol Res. 2006;55(5):513-526. doi: 10.33549/physiolres.930845. Epub 2005 Dec 12. PMID 16343035
- [Background] Ozkan G, Adar A, Ulusoy S, Bektas H, Kiris A, Fidan M, Celik S. Presence of fragmented QRS and its correlation with myocardial performance index in patients with nephrotic syndrome. Anadolu Kardiyol Derg. 2014 Aug;14(5):450-5. doi: 10.5152/akd.2014.4886. Epub 2014 Jan 28. PMID 24901023
- [Background] Loscalzo J. Venous thrombosis in the nephrotic syndrome. N Engl J Med. 2013 Mar 7;368(10):956-8. doi: 10.1056/NEJMcibr1209459. No abstract available. PMID 23465106